CLINICAL TRIAL: NCT05145387
Title: Transitioning Emotionally and Academically to Middle School Successfully: Development of a Brief Intervention to Reduce Student Anxiety (TEAMSS)
Brief Title: Transitioning Emotionally and Academically to Middle School Successfully (TEAMSS)
Acronym: TEAMSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-114-1; R324A200091 (Other Grant/Funding Number: Institution of Education Sciences)
Record Dates: First submitted 2021-11-05; First posted 2021-12-06 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Anxiety Disorders
Keywords: Middle school; Transition; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: independent evaluators
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAMSS Intervention in the RCT (Experimental): Students randomly assigned to the TEAMSS intervention will receive the 5th and 6th grade components.
  Interventions: Behavioral: Transitioning Emotionally and Academically to Middle School Successfully (TEAMSS)
- Enhanced Usual Care in the RCT (No Intervention): Enhanced Usual Care (EUC) will serve as the comparison group. EUC will be comprised of written materials (given all at once after randomization by study team) for parents and children that include: 1) a specialty mental health referral list; 2) a list of websites and books on child anxiety; and 3) tip sheets on successful transitions to MS. Families in this condition will not be prohibited from seeking treatment (though this will be monitored) for their children. These students will visit and meet with the 6th grade clinician in the spring of 5th grade.

INTERVENTIONS:
Behavioral: Transitioning Emotionally and Academically to Middle School Successfully (TEAMSS) — Students randomized to TEAMSS will receive reading materials on transitioning to middle school and a a school tour with the middle school clinician (in 5th grade) and the TEAMSS group sessions (in 6th grade) delivered over 10 weeks. During the 10 weeks of TEAMSS, parents of students will attend two group meetings and clinicians will consult with at least one teacher (usually the advisory/homeroom teacher).
  Arms: TEAMSS Intervention in the RCT

SUMMARY:
Excessive anxiety is a common problem that severely impairs short and long term academic functioning. The transition to middle school (MS) results in increases in anxiety and decreases in academic functioning. Students with anxiety in particular, due to their vulnerability to school-based stressors, are at risk for social, emotional and academic failure during the transition to MS. Unfortunately, the majority of these students do not get identified. Reducing student anxiety has been associated with improvement in academic functioning. Because the transition to MS is inevitable, targeting students with excessive anxiety will help their adjustment to their new school setting, reducing the need for special education and mental health counseling. No interventions exist to help these students with this transition.

This study aims to: (1) develop and assess the feasibility of a brief, multi-component intervention, referred to as TEAMSS, Transitioning Emotionally and Academically to Middle School Successfully, to reduce anxiety and improve academic functioning through the transition to MS using an iterative development process (i.e., expert review, two open trials, and small randomized controlled trial (RCT)); (2) conduct a pilot RCT comparing the preliminary impact of TEAMSS, relative to enhanced usual care (EUC), in improving students' social, behavioral, and academic functioning through the transition to MS; and (3) examine theory-based mediators, predictors, and moderators of TEAMSS and assess intervention costs.

DETAILED DESCRIPTION:
The pilot RCT will be conducted with approximately 8 school-based clinicians from 6-8 middles schools (MS). Approximately 42 5th grade students from 12 elementary schools with elevated anxiety will be recruited. The RCT will be conducted in 3 phases:

Phase 1 - Recruitment, Screening, Baseline Evaluation and Randomization: In Phase 1, 5th grade students will be referred to study staff for screening and evaluation from 5th grade teachers, clinicians and parents and self-referrals. Interested parents and students will contact study staff and complete a brief phone screen. Families who pass the screen will complete informed consent and the full baseline evaluation (consisting of a diagnostic interview and questionnaires) with an Independent Evaluator.

Phase 2 - Intervention and Monitoring: Eligible students will be randomized (1:1) to TEAMSS (n = 21) or Enhanced Usual Care (EUC; n= 21). Students in both groups will receive the 5th grade components but only students randomized to TEAMSS will receive the TEAMSS group sessions (in 6th grade), delivered over 10 weeks. During the 10 weeks of TEAMSS, parents of students will attend two group meetings and clinicians will consult with at least one MS teacher.

Phase 3 - Post- and Follow-up Evaluations: At the end of the 10-week intervention/EUC phase, students in both groups will complete the post-intervention (3 months into transition year i.e., December). Five months after the intervention ends (8 months into the transition year i.e., May), students in both groups will complete a follow up evaluation to assess the durability of the intervention. A seventh group with students, and a third group for parents, occurring approximately four weeks after session 6 will be conducted to debrief (discuss their experience in the program), ask them about any lingering questions or concerns related to anxiety, and update them on what was learned.

ELIGIBILITY:
Student:

Inclusion Criteria:

* be in the last year of a participating elementary school
* have elevated anxiety symptoms that are their primary concern as indicated by 1) a total SCARED score at baseline of 15 or higher using parent and/or child report, and/or 2) a Clinician Severity Rating (CSR) of 3 or higher on the ADIS
* read and understand English (both parent and child).

Exclusion Criteria:

* Students who have a non-anxiety primary mental health concern (e.g., ADHD) will be excluded from TEAMSS, as this intervention is aimed at reducing anxiety and it would not be effective at treating other mental health concerns. Students with comorbid conditions secondary to anxiety will be eligible.

Clinician:

Inclusion Criteria:

* All clinician participants must be at least a part time employee of a CT MS in the role of school clinician.

Exclusion Criteria:

* None

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Global Impression - Severity (CGI-S) Scale | Change from baseline (before intervention) to follow up at 8 months
  The CGI-S score provides a global rating of anxiety severity ranging from 1= "not at all ill" to 7= "extremely ill".
Change in Clinical Global Impression - Improvement (CGI-I) Scale | Change from post intervention evaluation to follow up at 8 months
  The CGI-I provides a global rating of clinical improvement in anxiety (relative to baseline) ranging from 1= "very much improved" to 7= "very much worse." Scores of 1-2 are considered "responders."

SECONDARY OUTCOMES:
Change in Screen for Child Anxiety Related Emotional Disorders, Child and Parent Versions (SCARED) | Change from baseline (before intervention) to follow up at 8 months
  A widely used 41 item measure of childhood anxiety. Informants respond to items using a 3-point Likert-type scale (0 = "not true or hardly ever true", 1 = "somewhat true or sometimes true", 2 = "very true or often true").
Change in Anxiety Disorders Interview Schedule for DSM-V, Parent and Child Versions (ADIS-V) | Change from baseline (before intervention) to follow up at 8 months
  Considered the gold standard for assessing anxiety diagnosis and severity. Impairment ratings are generated for each disorder using the Clinician Severity Rating (CSR, range = 0-8; 4 or higher is required to assign a diagnosis).
Change in Child Anxiety Impact Scale (CAIS) | Change from baseline (before intervention) to follow up at 8 months
  A 27 item measure of anxiety-related interference in social, academic and family functioning. It is scored on a 4-point Likert scale, from 0= "not at all" to 3= "very much."
Change in School Anxiety Scale - Teacher Report (SAS) | Change from baseline (before intervention) to follow up at 8 months
  The SAS is a 16 item questionnaire of student anxiety, items are rated on a 3 point scale (0 = "never" to 3 = "always").
Change in School Records | Change from baseline (before intervention) to follow up at 8 months
  Assess grades, attendance, referrals for special education, grade retention and referrals for disciplinary actions (e.g., suspensions, detentions).
Change in Academic Competence Evaluation Scale (ACES) | Change from baseline (before intervention) to follow up at 8 months
  A 50 item questionnaire, scored on a 5-point Likert scale ranging from "never" to "almost always" that assesses: Academic Skills (reading, mathematics, critical thinking) and Academic Enablers (Motivation, Engagement, Study Skills, Interpersonal Skills).
Change in Subtests from the Woodcock-Johnson IV Tests of Achievement and Cognitive Abilities (WJ IV) | Change from baseline (before intervention) to follow up at 8 months
  These subtests are a widely used, norm-referenced measure of academic achievement and cognitive abilities. Reading, math fluency and numbers reversed will be administered to measure cognitive factors (e.g., efficiency, speed, working memory) that are affected by anxiety.
Change in Children's Automatic Thoughts Scale (CATS) | Change from baseline (before intervention) to follow up at 8 months
  A 40 item questionnaire of maladaptive thoughts associated with anxiety. Items are scored on a 5-point Likert scale from 0= "not at all" to 4= "all the time." To reduce burden, only the Physical and Social Threat subscale will be used.
Change in Avoidance Hierarchy | Change from baseline (before intervention) to follow up at 8 months
  A 3 item measure used in our ongoing studies, which assesses how frequently the student avoids specific anxiety provoking situations from 1 = "never" to 7 = "every time."
Change in Children's Somatization Inventory (CSI-24) | Change from baseline (before intervention) to follow up at 8 months
  A 24 item measure of the child's somatic symptoms (headaches, stomach aches). Items are ranked using a 5 point scale ranging from "not at all" to "a whole lot."
Change in My Memories of Growing Up (Egna Minnen Beträffande Uppfostran; EMBU) | Change from baseline (before intervention) to follow up at 8 months
  A 40 item measure of parental over control and anxious rearing practices associated with higher anxiety. This scale consists of four subscales with 10 items each: overprotection/control, emotional warmth, rejection, and anxious rearing. For purposes of this study, only the overprotection/control and anxious rearing subscales will be used. Items are answered on a 4-point Likert scale ranging from 1= "no," to 4= "yes, most of the time."
Change in Family Accommodation Scale - Anxiety (FASA) | Change from baseline (before intervention) to follow up at 8 months
  A measure of accommodation. Parents respond to 9 items, which are coded on a 5-point Likert scale from 0 = "never" to 4 = "daily."
Change in Children's Organizational Skills Scale (COSS) | Change from baseline (before intervention) to follow up at 8 months
  A 41 item parent, teacher and child measure of organization, planning and time-management. The COSS yields three subscale scores: task planning, organized actions and memory and materials management.
Change in Children's Global Assessment Scale (CGA-S) | Change from baseline (before intervention) to follow up at 8 months
  A measure to assess the student's overall improvement, as a result of participating in the intervention.
Change in Strength and Difficulties Questionnaire Parent Version (SDQ | Change from baseline (before intervention) to follow up at 8 months
  A widely used and psychometrically sound (alpha = .80) 25 item parent report questionnaire that assesses emotional and behavioral difficulties in children 4-17 years old. It yields a total score and five subscale scores: emotion problems, conduct problems, hyperactivity, peer problems and prosocial.
Change in Revised Child Anxiety and Depression Scale - Depression subscale only (RCADS) | Change from baseline (before intervention) to follow up at 8 months
  The RCADS Depression subscale is comprised of 10 items. Youth respond to items using a 4-point Likert-type scale (0-3) to indicate the frequency of symptoms: 'never,' 'sometimes,' 'often,' and 'always.' Higher scores reflect greater frequency of depressive symptoms.

OTHER OUTCOMES:
Change in TEAMSS Intervention Satisfaction Questionnaire | Change from post intervention evaluation to follow up at 8 months
  This measure will be modified from the PI's studies (Ginsburg et al., 2019a).
Change in The Child and Adolescent Services Assessment (CASA) | Change from baseline (before intervention) to follow up at 8 months
  A 20-item measure assessing the use of general medical health, mental health, social service, and education services. Items are rated on a yes/no scale. The measure includes checkboxes for participants to indicate details about the services (e.g., frequency, indication, provider).

CONTACTS AND LOCATIONS:
Overall Officials: Golda Ginsburg, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT05145387/ICF_000.pdf